CLINICAL TRIAL: NCT05221944
Title: Perioperative Safety of Bladder Hydrodistension in Patients on Antithrombotic Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, De-yi Luo, Prof., West China Hospital
Other Study IDs: 2019186
Record Dates: First submitted 2022-01-04; First posted 2022-02-03 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Complication
Keywords: Interstitial cystitis; Antithrombotic therapy; Complication; Bladder hydrodistension
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients on antithrombotic therapy: The study aimed to investigate if perioperative bleeding complications were more common in patients on antithrombotic therapy. We retrospectively reviewed patients with IC/BPS who underwent hydrodistension during January 2010 and May 2021. Patients with and without antithrombotic drugs were identified and grouped and their medical records were reviewed.
  Interventions: Other: Patients had a history of antithrombotic therapy
- Patients without antithrombotic therapy: Patients without antithrombotic drugs were identified as controls
  Interventions: Other: Patients had no history of antithrombotic therapy

INTERVENTIONS:
Other: Patients had a history of antithrombotic therapy — Patients with antithrombotic drugs were identified and grouped and their medical records were reviewed.
  Groups: Patients on antithrombotic therapy
Other: Patients had no history of antithrombotic therapy — Patients had no history of antithrombotic therapy
  Groups: Patients without antithrombotic therapy

SUMMARY:
After obtaining an institutional ethics approval (#2019186), we retrospectively reviewed patients with interstitial cystitis/bladder pain syndrome (IC/BPS) who underwent hydrodistension in our hospital during January 2010 and May 2021. The diagnosis of IC/BPS was made by the same senior urologist according to the National Institute of Diabetes, Digestive and Kidney Diseases guidelines. Patients who met the inclusion and exclusion criteria were considered eligible for the study. Medical records were reviewed to extract baseline information, including age, body mass index (BMI), duration, antithrombotic use and classification, symptom assessment, and perioperative parameters. Patients were then contacted and volunteered to undergo a follow-up. Telemedicine-based follow-ups were performed at 3 after surgery. Complications and symptoms were recroded. Then, perioperative parameters, including operation time, hospital stays, catheterization time, and hematological results (hemoglobin, platelet count, and coagulated parameters) were recorded based on medical records. The data were analyzed to investigate if perioperative complications were more common in patients with IC/BPS on antithrombotic therapy after bladder hydrodistension.

DETAILED DESCRIPTION:
Study population. This retrospective study was performed in line with STROCSS guidelines. After obtaining an institutional ethics approval (#2019186), we retrospectively reviewed patients with IC/BPS who underwent hydrodistension in our hospital during January 2010 and May 2021. The diagnosis of IC/BPS was made by the same senior urologist according to the National Institute of Diabetes, Digestive and Kidney Diseases guidelines. A stepwise procedure of elimination of disorders with similar symptoms was performed. Generally, urinalysis and urine culture were performed to exclude UTI and some specific infections, ultrasound and imaging were conducted to exclude malformation, carcinoma and urinary stones, and urodynamic studies were performed to assess functional disorders. Patients who met the inclusion and exclusion criteria were considered eligible for the study. Medical records were reviewed to extract baseline information, including age, body mass index (BMI), duration, antithrombotic use and classification, symptom assessment, and perioperative parameters. Patients were then contacted and volunteered to undergo a follow-up.

Antithrombotic therapy. Antithrombotic drugs in the current study included anticoagulation (heparin, warfarin, as well as rivaroxaban) and antiplatelet drugs (aspirin, clopidogrel). The study aimed to investigate if perioperative bleeding complications were more common in patients on antithrombotic therapy. The algorithm of managing antithrombotic use is based on clinical practice. After a cardiologic and anesthetic consultation, patients taking aspirin remained on therapy throughout the procedure and after the procedure. Clopidogrel was held 5 days before hydrodistension and was restarted 24 hours postoperatively. Both low molecular weight heparin (LMWH) and rivaroxaban were discontinued 1 day before surgery and were restarted one day postoperatively. Warfarin was held 5 days before hydrodistension and was restarted 12 hours postoperatively, keeping an international normalized ratio (INR) 2-3.

Bladder hydrodistension. All patients signed informed consents. Patients' basic conditions were carefully evaluated and managed before surgery. The hydrodistension was in a day-surgery setting in our institute and was performed by the same urologist or under his supervision. Broad spectrum antibiotics were given 30 minutes preoperatively. After general anesthesia, Hunner lesions were identified by cystoscopy with the bladder slightly filled with saline. Then, the bladder was distended with normal saline at the pressure of 70 cmH2O for 2 minutes. Under this circumstance, a waterfall bleeding sign from Hunner lesion or glomerulations in submucosa might be visualized. Subsequently, biopsy was performed to exclude carcinomas in situ. At last, a 16 Fr three-way catheter was inserted with continuous saline irrigation. The time to remove catheters and the time to discharge after voiding tests were decided by the treating physician. Intravesical instillation of hyaluronic acid was performed as a follow-up treatment for all patients according to the instructions. Telemedicine-based follow-ups were performed at 3 months after surgery. Perioperative parameters, including operation time, hospital stays, catheterization time, and hematological results (hemoglobin, platelet count, and coagulated parameters) were recorded.

Outcomes. Primary outcomes were complications that were defined by Clavien-Dindo classification of surgical complications. The complications were recoded within 3 months after surgery. Then, the mean frequency of voids per day, number of night urination, O'Leary-Sant Interstitial Cystitis Symptom index (ICSI), O'Leary-Sant Interstitial Cystitis Problem Index (ICPI), and 10-point visual analog scale (VAS) 3 months postoperatively were analyzed to evaluate the improvement of symptoms.

Data analysis. SPSS software (version 25) and GraphPad Prism software (version 8.0) were applied to perform all statistical analyses. Continuous variables are presented as the means ± standard deviation or medians (range), and differences between groups were tested using the Student's t test or the Mann-Whitney U test, respectively. The changes of pre- and postoperative continuous variables were tested by the paired t test. Categorical parameters were reported as the numbers (percentage), and the chi-square test with and without Yates' correction was applied where appropriate. Subsequently, odd ratio (OR) and 95% confidence interval of each adverse event after antithrombotic use were calculated. A p value of < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old when signing an informed consent;
2. Previously diagnosed with IC/BPS for a duration of > 6 months;
3. O'Leary-Sant Interstitial Cystitis Symptom and Problem Index scores over 18;
4. Undergoing hydrodistension during the hospitalization;
5. Patients with adequate medical records.

Exclusion Criteria:

1. General conditions 1) Currently diagnosed with cancer, or have previous history of cancer within the preceding 5 years; 2) Currently diagnosed with severe heart, lung, liver, kidney, or blood disorders; 3) Pregnant women.
2. Urological symptoms 1) Have previous history of urinary infection (e.g., bacterial cystitis, bladder tuberculosis, urethritis, genital chlamydia infection, and genital herpes) within 12 weeks; 2) Currently diagnosed with any of following diseases, which had similar symptoms with IC/BPS.

   1. Bladder diseases (carcinoma, overactive bladder, neurogenic bladder, bladder stone, radiation cystitis)
   2. Urethral diseases (urethral diverticulum, urethral stricture, urethral stone)
   3. Gynaecological diseases (endometriosis, uterine fibroids, vaginitis, menopausal syndrome, pelvic organ prolapse)
   4. Others (neurogenic urinary frequency, polyuria) 3) Have previous history of augmentation cystoplasty or cystectomy; 4) Have previous history of chemical compound (such as cyclophosphamide) derived cystitis.
3. Treatment related 1) History of the following therapies within 12 weeks: hydrodistension, intravesical laser therapy, intravesical electrical coagulation, transurethral resection, pelvic reconstructive surgery, nerve stimulation for pain relief; 2) Received intravesical instillation of any drugs within 12 weeks.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: After obtaining an institutional ethics approval (#2019186), we retrospectively reviewed patients with IC/BPS who underwent hydrodistension in our hospital during January 2010 and May 2021. The diagnosis of IC/BPS was made by the same senior urologist according to the National Institute of Diabetes, Digestive and Kidney Diseases guidelines. A stepwise procedure of elimination of disorders with similar symptoms was performed. Patients who met the inclusion and exclusion criteria were considered eligible for the study. Medical records were reviewed to extract baseline information, including age, body mass index (BMI), duration, antithrombotic use and classification, symptom assessment, and perioperative parameters. Patients were then contacted and volunteered to undergo a follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 387 (Estimated)
Dates: Start 2019-07-04 (Actual); Primary Completion 2024-02-10 (Estimated); Study Completion 2024-04-10 (Estimated)

PRIMARY OUTCOMES:
Complications | The complications were recoded within 3 months after surgery.
  Primary outcomes were complications that were defined by Clavien-Dindo classification of surgical complications.

SECONDARY OUTCOMES:
The mean frequency of voids per day | The data were recoded at 3 months after surgery.
  Change from baseline voids at 3 months.
The mean number of night urination | The data were recoded at 3 months after surgery.
  Change from baseline night urination at 3 months.
O'Leary-Sant Interstitial Cystitis Symptom index (0-19). Higher scores mean a worse outcome. | The data were recoded at 3 months after surgery.
  Change from baseline symptom index at 3 months.
O'Leary-Sant Interstitial Cystitis Problem Index (0-16). Higher scores mean a worse outcome. | The data were recoded at 3 months after surgery.
  Change from baseline problem index at 3 months.
Visual analog scale (0-10). Higher scores mean a worse outcome. | The data were recoded at 3 months after surgery.
  Change from baseline pain index at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-min Li, PhD., Study Chair — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided